CLINICAL TRIAL: NCT02877056
Title: Molecular Determinants of Response to Preoperative Therapy in Patients With Locally Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Research Foundation of the American Society of Colon and Rectal Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: LAB04-0962; R33 CA118505-01 (Other Grant/Funding Number: American Society of Colon and Rectal Surgeons Research)
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal adenocarcinoma; Neoadjuvant therapy; Endoscopy; Endoscopic biopsy; Biomarkers; Genes
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples taken from tumor and normal colorectal tissue during standard endoscopy.
  Up to eight biopsy samples of the tumor as well as up to six biopsies of the grossly normal colorectum obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Cancer: Participants undergo standard endoscopy before therapy. Tissue samples taken from the tumor and normal colorectal tissue.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Tissue samples taken from tumor and normal colorectal tissue during standard endoscopy before therapy.

SUMMARY:
The goal of this laboratory research is to look for genes that can predict which patients will achieve a complete disappearance of their colorectal cancer after treatment like chemotherapy, radiation, or other therapy.

This is an investigational study. Up to 350 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Patients with colorectal cancer usually receive radiation, chemotherapy, or other therapy before they have surgery. At this time, there are no tests that can help researchers find out which patients no longer have any tumor left after completing treatment. Because of this, all patients have to have surgery to completely remove the rectum and/or part of the colon. This procedure results in lifestyle changes for the patient, which may be difficult and permanent.

Researchers are looking for new ways to find out which patients will have no tumor left after treatment, so that in the future, some patients may be able to avoid surgery altogether. In this study, researchers will try to use chemical "markers" in tumor cells as a way to possibly predict whether or not the tumor is likely to disappear with treatment alone.

At MD Anderson, all patients with colorectal cancer have an endoscopy performed by their surgeon as part of standard care, before they start therapy. Endoscopy involves placing a narrow tube in the colon and/or rectum in order to see and inspect the tumor.

If you choose to take part in this study, tissue samples will be taken from the tumor and the normal areas during your standard endoscopy. If you undergo surgery, tissue samples from the tumor(s) and normal areas will also be collected. At the time of endoscopy and/or surgery, once the doctor has finished all standard tests on this tissue and has received the clinical reports on these tests, any leftover tissue samples will be collected by Dr. You or a person on her research team for research tests to look for tumor cell "markers." Researchers want to find out how these markers may have changed since you began receiving treatment for the disease.

Some of the tissue from your biopsies may also be sent to the labs at University of Texas-Southwest or Natera for testing. No identifying information about you will be included with these samples. They will have a special number assigned, so that the samples being sent to UT Southwest or Natera will not be able to be connected to you in any way.

The results of these tests will not be used to make any decisions regarding treatment of your rectal cancer. There are no other tests or procedures required in this study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal adenocarcinoma (diagnosis based on either MDACC or outside records)
2. Patients scheduled to undergo neoadjuvant therapy per MDACC care team.
3. Patients over 18 years of age.
4. Patients with distant organ findings deemed to be indeterminate or metastatic will be enrolled at the surgeon's discretion.
5. Patients who have been deemed medically safe to undergo endoscopic biopsy by the physician performing the procedure.
6. Patients who would have typically undergone preoperative therapy followed by surgery but for specific reasons at the discretion of the treating physician underwent surgery without preoperative therapy may be enrolled at the surgeons' discretion.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Colorectal Cancer in the Gastrointestinal (GI) department at University of Texas MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Predictive Tumor Cell Biomarkers After Chemoradiation Treatment for Colorectal Cancer | 1 day
  Tissue taken at endoscopy undergoes testing for tumor cell biomarkers to identify patients who achieve complete response (CR).

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Qian N. You, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org